CLINICAL TRIAL: NCT04600739
Title: Entscheidungsunterstützung Bei Herzklappenerkrankungen Anhand Funktionaler Und Morphologischer Eigenschaften Mittels Methoden Der Mathematischen Modellierung Und Des Maschinellen Lernens
Brief Title: Validation of a Novel, Non-Dimensional Approach for Estimation of Pressure Gradients in Aortic Stenosis
Acronym: AVD-PowerLaw
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: German Heart Institute (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Other Study IDs: AVD-PowerLaw
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AVD Patients: Patients suffering from aortic valve stenosis receiving replacement of the diseased valve using a TAVI procedure.
  Interventions: Procedure: TAVI

INTERVENTIONS:
Procedure: TAVI — Replacement of the aortic valve using a biological prosthesis that is inserted via a catheter.

SUMMARY:
A novel, image-based model for estimation of the pressure gradient across stenosed aortic valves is compared against invasively measured pressure gradients from clinical routine.

DETAILED DESCRIPTION:
Using temporally resolved computed tomography images, the patient-specific geometry of the stenosed aortic valve during peak systole is reconstructed. Using this geometry, the projected area of the aortic valve's orifice (AVA) is calculated. Additionally, the left ventricular geometry is reconstructed for the complete heart cycle. Using the information of the left ventricular volume change, the patient-specific flow profile and peak-systolic flow (Q)is calculated. Using this information, the pressure gradient is calculated using a power law estimation of the form PG = a * AVA^b * Q^c. The model generation and parameter fit is described in [1].

To validate this model, retrospective data of patients receiving a catheter-based replacement of the aortic valve (TAVI) is collected. For those patients, CT images are already acquired for treatment planning and the invasive pressure measurements are performed during replacement of the aortic valve. Therefore, no additionally steps are required. Using the CT images the patient-specific aortic valve area ad flow rate are calculated. This information is then used for estimation of the pressure gradient using the power law model. The catheter-based pressure gradient is calculated as the difference between the peak-systolic pressure in the left ventricle and the ascending aorta before implantation of the prosthesis.

[1] Franke et al.; Towards improving the accuracy of aortic transvalvular pressure gradients: rethinking Bernoulli; Medical & Biological Engineering & Computing (2020); https://doi.org/10.1007/s11517-020-02186-w

ELIGIBILITY:
Inclusion Criteria:

* aortic valve stenosis
* treatment via TAVI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: - retrospective acquisition of patients that receive TAVI
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
predicted vs. cather-measured pressure gradient across the aortic valv | 1 week up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Deutsches Herzzemtrum Berlin, Berlin, Deutschland, Germany

IPD SHARING:
Plan to Share IPD: No